CLINICAL TRIAL: NCT05566197
Title: Nusantara Diet (Balance Nutrition With Low Calorie and Low Sodium Diet) Impact on Body Composition, Insulin Resistance, and Lipid Profile in Patients With Risk of Metabolic Syndrome
Brief Title: Nusantara Diet (Low Calorie and Low Sodium) for Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0709221426
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Metabolic Syndrome; Diabetes; Hyperlipidemias
Keywords: Diet Nusantara; Low Calorie; Low Sodium; Lipid Profile; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Hyperlipidemias; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: The intervention will receive a package of dietary intervention + nutrition counseling, whereas the control group will receive only nutrition counseling.
Masking Description: masking is not feasible according to the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive dietary adjustment and nutrition counseling.
  Interventions: Dietary Supplement: Diet Nusantara; Behavioral: Nutrition Counseling
- Control (Active Comparator): This group will receive standard diet and nutrition counseling.
  Interventions: Behavioral: Nutrition Counseling

INTERVENTIONS:
Dietary Supplement: Diet Nusantara — Diet Nusantara consists of 1700 kilocalories (or 500 kilocalories lower than basal energy expenditure) on first month and subsequent reduction for the following months (200 kilocalories). The participants should also limit the sodium intake not more than 2300 mg daily
  Arms: Intervention
Behavioral: Nutrition Counseling — Nutrition counseling consists of the definition of balancing food, metabolic syndrome, exercise, and related health parameters.

SUMMARY:
The goal of this randomized clinical trial is to evaluate the effect of Nusantara Diet (Low Calorie and Low Sodium) for Metabolic Syndrome. The main questions it aims to answer are:

* How effective the Nusantara diet in reducing body mass index and body fat percentage?
* How effective the Nusantara diet in affecting lipid profile and insulin resistance?

Participants will be given this diet for a period of 56 days and undergo repeated outcome measurement. This study has a comparison group (no intervention) to see the difference of reduction or slope of changes in outcomes. We assumed that the Nusantara diet will reduce the metabolic syndrome indicators (anthropometry, lipid profile, and insulin resistance profile).

DETAILED DESCRIPTION:
Design

a. Randomized controlled trial with pre-post design

Intervention :

1. Balance Nutrition with low calorie and low sodium. Low calorie means a diet with 500 kilocalories lower than the Basal Energy Expenditure, according to the Harris-Benedict formula. The daily limit of sodium is 2300 mg.
2. Organoleptic test for set menu
3. Given as a set for 56 days
4. Dietary counseling is given before intervention, followed by a 24-hour food recall every week.

Outcome

1. Body mass index
2. Blood chemistry test: Total Cholesterol, Low-Density Lipoprotein (LDL), High-density Lipoprotein, Triglyceride,

4. Glucose profile (Fasting blood glucose, and Homeostatic Model Assessment for Insulin Resistance / HOMA-IR) 3. Body Fat percentage using Bioelectrical Impedance Analyzer

Sample Size Estimation With the following assumption

1. Type I error: 5%
2. Power of Study: 80%
3. Superiority Trial
4. Equal allocation with two arms
5. Assuming that the reduction of LDL would be 30% of the average LDL level among metabolic syndrome individuals (106.4 mg/dL), the total sample would be 48 participants

Protocol Analysis

1. Intention-to-treat analysis
2. Sensitivity analysis and subgroup analysis
3. If the randomization obtains an equal baseline characteristic, an Independent T-test will be applied.
4. Regression model will be applied, adjusting any possible confounder.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the definition of metabolic syndrome

  1. Blood Pressure>135/85 mmHg
  2. Central obesity with waist circumference for males>90 cm or >80 cm in females
  3. Triglyceride level >150 mg/dL, followed by HDL<40 mg/dL
  4. blood fasting glucose >100 mg/dL

Exclusion Criteria:

1. pregnant or breastfeeding women
2. suffer from chronic disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | changes of body mass index from baseline to day 56
  Defined as body weight in kilogram defined by square of body height in meter. Higher number indicates obesity
Lipid profile | changes of lipid profile from baseline to day 56
  parameters of lipid (total cholesterol, LDL, HDL, Triglyceride) measured from blood sample
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | changes of HOMA-IR from baseline to day 56
  HOMA-IR was calculated according to the formula: fasting insulin x fasting glucose/22.5.
Body Fat Percentage | changes of Body Fat Percentage from baseline to day 56
  Body Fat Percentage is the total mass of fat divided by total body mass, multiplied by 100. This is measured by Bioelectrical Impedance Analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Agussalim Bukhari, MD.Phd, Principal Investigator — Hasanuddin University
Locations (1):
- Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
De-identified data in a form of publication supplement will be shared accordingly

REFERENCES:
- [Background] Sigit FS, Tahapary DL, Trompet S, Sartono E, Willems van Dijk K, Rosendaal FR, de Mutsert R. The prevalence of metabolic syndrome and its association with body fat distribution in middle-aged individuals from Indonesia and the Netherlands: a cross-sectional analysis of two population-based studies. Diabetol Metab Syndr. 2020 Jan 7;12:2. doi: 10.1186/s13098-019-0503-1. eCollection 2020. PMID 31921359
- [Background] Rochlani Y, Pothineni NV, Kovelamudi S, Mehta JL. Metabolic syndrome: pathophysiology, management, and modulation by natural compounds. Ther Adv Cardiovasc Dis. 2017 Aug;11(8):215-225. doi: 10.1177/1753944717711379. Epub 2017 Jun 22. PMID 28639538
- [Background] Papamandjaris AA, MacDougall DE, Jones PJ. Medium chain fatty acid metabolism and energy expenditure: obesity treatment implications. Life Sci. 1998;62(14):1203-15. doi: 10.1016/s0024-3205(97)01143-0. PMID 9570335
- [Background] Lipoeto NI, Agus Z, Oenzil F, Wahlqvist M, Wattanapenpaiboon N. Dietary intake and the risk of coronary heart disease among the coconut-consuming Minangkabau in West Sumatra, Indonesia. Asia Pac J Clin Nutr. 2004;13(4):377-84. PMID 15563444
- [Background] de la Iglesia R, Loria-Kohen V, Zulet MA, Martinez JA, Reglero G, Ramirez de Molina A. Dietary Strategies Implicated in the Prevention and Treatment of Metabolic Syndrome. Int J Mol Sci. 2016 Nov 10;17(11):1877. doi: 10.3390/ijms17111877. PMID 27834920
- [Background] Goossens GH. The Metabolic Phenotype in Obesity: Fat Mass, Body Fat Distribution, and Adipose Tissue Function. Obes Facts. 2017;10(3):207-215. doi: 10.1159/000471488. Epub 2017 Jun 1. PMID 28564650
- [Background] Di Daniele N, Noce A, Vidiri MF, Moriconi E, Marrone G, Annicchiarico-Petruzzelli M, D'Urso G, Tesauro M, Rovella V, De Lorenzo A. Impact of Mediterranean diet on metabolic syndrome, cancer and longevity. Oncotarget. 2017 Jan 31;8(5):8947-8979. doi: 10.18632/oncotarget.13553. PMID 27894098
- [Background] Gusnedi, Abdullah M, Witjaksono F, Mansyur M, Nurwidya F, Djuwita R, Dwiriani CM, Fahmida U. Promotion of optimized food-based recommendations to improve dietary practices and nutrient intakes among Minangkabau women of reproductive age with dyslipidemia. Asia Pac J Clin Nutr. 2020;29(2):334-347. doi: 10.6133/apjcn.202007_29(2).0016. PMID 32674241